CLINICAL TRIAL: NCT03249376
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Assess the Efficacy and Safety of Lumateperone Monotherapy in the Treatment of Patients With Major Depressive Episodes Associated With Bipolar I or Bipolar II Disorder (Bipolar Depression) Conducted Globally
Brief Title: Lumateperone Monotherapy for the Treatment of Bipolar Depression Conducted Globally
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITI-007-404
Record Dates: First submitted 2017-08-11; First posted 2017-08-15 (Actual); Results first posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — lumateperone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lumateperone (Experimental): Lumateperone 42 mg (ITI-007 60 mg tosylate) administered once daily every evening for 6 weeks
  Interventions: Drug: Lumateperone
- Placebo (Placebo Comparator): Placebo administered once daily every evening for 6 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lumateperone — Lumateperone 42 mg (ITI-007 60 mg tosylate)
  Other Names: ITI-007
  Arms: Lumateperone
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The study will evaluate the efficacy and safety of ITI-007 in a randomized, double-blind, parallel-group, placebo-controlled, multi-center study in patients diagnosed with Bipolar I or Bipolar II disorder having a major depressive episode.

ELIGIBILITY:
Major Inclusion Criteria:

* male or female subjects of any race, ages 18-75 inclusive, with a clinical diagnosis of Bipolar I or Bipolar II disorder
* experiencing a current major depressive episode
* able to provide written informed consent

Major Exclusion Criteria:

* any female subject who is pregnant or breast-feeding
* any subject judged to be medically inappropriate for study participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Kozauer, MD, Study Director — Intra-Cellular Therapies, Inc.
Locations (47):
- United States (14):
  - Clinical Site, Birmingham, Alabama
  - Clinical Site, Sherman Oaks, California
  - Clinical Site, Miami, Florida
  - Clinical Site, Orange City, Florida
  - Clinical Site, Atlanta, Georgia
  - Clinical Site, Decatur, Georgia
  - Clinical Site, Chicago, Illinois
  - Clinical Site, Joliet, Illinois
  - Clinical Site, Shreveport, Louisiana
  - Clinical Site, St Louis, Missouri
  - Clinical Site, Buffalo, New York
  - Clinical Site, Charlotte, North Carolina
  - Clinical Site, The Woodlands, Texas
  - Clinical Site, Bothell, Washington
- Bulgaria (10):
  - Clinical Site, Burgas
  - Clinical Site, Kardzhali
  - Clinical Site, Lovech
  - Clinical Site, Plovdiv
  - Clinical Site, Rousse
  - Clinical Site, Sofia
  - Clinical Site, Targovishte
  - Clinical Site, Tsarev Brod
  - Clinical Site, Varna
  - Clinical Site, Veliko Tarnovo
- Colombia (3):
  - Clinical Site, Barranquilla
  - Clinical Site, Bello
  - Clinical Site, Pereira
- Russia (8):
  - Clinical Site, Moscow
  - Clinical Site, Nizhny Novgorod
  - Clinical Site, Omsk
  - Clinical Site, Saint Petersburg
  - Clinical Site, Samara
  - Clinical Site, Saratov
  - Clinical Site, Tomsk
  - Clinical Site, Yekaterinburg
- Serbia (3):
  - Clinical Site, Belgrade
  - Clinical Site, Kragujevac
  - Clinical Site, Novi Sad
- Ukraine (9):
  - Clinical Site, Ivano-Frankivsk
  - Clinical Site, Kharkiv
  - Clinical Site, Kherson
  - Clinical Site, Lviv
  - Clinical Site, Odesa
  - Clinical Site, Poltava
  - Clinical Site, Smila
  - Clinical Site, Uzhhorod
  - Clinical Site, Vinnytsia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] McIntyre RS, Durgam S, Huo J, Kozauer SG, Stahl SM. The Efficacy of Lumateperone in Patients With Bipolar Depression With Mixed Features. J Clin Psychiatry. 2023 Apr 24;84(3):22m14739. doi: 10.4088/JCP.22m14739. PMID 37103915
- [Derived] Calabrese JR, Durgam S, Satlin A, Vanover KE, Davis RE, Chen R, Kozauer SG, Mates S, Sachs GS. Efficacy and Safety of Lumateperone for Major Depressive Episodes Associated With Bipolar I or Bipolar II Disorder: A Phase 3 Randomized Placebo-Controlled Trial. Am J Psychiatry. 2021 Dec;178(12):1098-1106. doi: 10.1176/appi.ajp.2021.20091339. Epub 2021 Sep 23. PMID 34551584

RESULTS

PARTICIPANT FLOW:
Groups:
- Lumateperone: Lumateperone 42 mg (ITI-007 60 mg tosylate) administered once daily every evening for 6 weeks
  Lumateperone: Lumateperone (ITI-007 60 mg tosylate)
Period: Overall Study
Arm/Group | Lumateperone | Placebo
Started | 188 (191 patients were randomized but only 188 patients received study drug. The number completed and discontinued is based on the 188 patients that received study drug.) | 189 (190 patients were randomized but only 189 patients received study drug. The number completed and discontinued is based on the 189 patients that received study drug.)
Completed | 167 | 166
Not Completed | 21 | 23
Not completed — Adverse Event | 11 | 5
Not completed — Lack of Efficacy | 2 | 4
Not completed — Protocol Violation | 3 | 2
Not completed — Physician Decision | 0 | 2
Not completed — Withdrawal by Subject | 3 | 9
Not completed — LTFU | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lumateperone | Placebo | Total
Number analyzed (Participants) | 188 | 189 | 377
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (14.09) | 44.1 (12.87) | 44.9 (13.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 120 | 219
  Male | 89 | 69 | 158
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White | 173 | 171 | 344
  Black or African American | 14 | 15 | 29
  Asian | 1 | 0 | 1
  Other | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 51 | 59 | 110
  Ukraine | 49 | 38 | 87
  Bulgaria | 49 | 43 | 92
  Serbia | 6 | 13 | 19
  Russia | 32 | 34 | 66
  Colombia | 1 | 2 | 3
Montgomery-Asberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: units on a scale] — The Montgomery-Åsberg Depression Rating Scale (MADRS) is a clinician-rated 10 item scale to assess depressive symptoms. Each item is rated on a 7-point scale from 0-6. The total score ranges from 0 to 60 with a higher score indicating increased severity of depressive symptoms.
  units on a scale | 30.8 (4.92) | 30.2 (4.65) | 30.5 (4.79)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score
Description: The Montgomery-Åsberg Depression Rating Scale (MADRS) is a clinician-rated 10 item scale to assess depressive symptoms. Each item is rated on a 7-point scale from 0-6. The total score ranges from 0 to 60 with a higher score indicating increased severity of depressive symptoms.
Time Frame: Baseline to Day 43
Population: Intent-to-Treat (ITT) Set contains all randomized patients who received at least one dose of study medication and had a valid baseline (pre-dose) measurement and at least one valid post-baseline measurement of MADRS total score.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Lumateperone | Placebo
Number analyzed (Participants) | 188 | 188
score on a scale | -16.70 (0.693) | -12.12 (0.677)
Statistical Analysis 1: Comparison: Lumateperone vs Placebo; Test type: Superiority; p < 0.0001, Mixed Effects Model for Repeated Measure; Least Squares Mean Difference = -4.6, 95% CI 2-sided [-6.34 to -2.83], Standard Error of Mean 0.89

2. Secondary Outcome: Change From Baseline in Clinical Global Impression Scale, Bipolar Version (CGI-BP-S) Total Score
Description: The Clinical Global Impression Scale, Bipolar version (CGI-BP-S) total score is a clinician-rated scale that measures the patient's current illness state on a 3 to 21 point scale where a higher score is associated with greater illness severity.. Each domain (depression, mania, and overall illness) is rated from 1 (not ill at all) to 7 (among the most extremely ill) and the 3 scores are added to obtain the total score.
Time Frame: Baseline to Day 43
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Lumateperone | Placebo
Number analyzed (Participants) | 188 | 188
score on a scale | -3.48 (0.170) | -2.54 (0.167)
Statistical Analysis 1: Comparison: Lumateperone vs Placebo; Test type: Superiority; p < 0.0001, Mixed Effects Model for Repeated Measure; Least Squares Mean Difference = -0.9, 95% CI 2-sided [-1.37 to -0.51], Standard Error of Mean 0.22

3. Secondary Outcome: Change From Baseline in Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) Percent Score
Description: The Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) is a 14 item patient self-reported questionnaire that assesses how satisfied a patient is, using a 5-point scale from 1-very poor to 5-very good.
Time Frame: Baseline to Day 43
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent Score
Arm/Group | Lumateperone | Placebo
Number analyzed (Participants) | 188 | 188
Percent Score | 19.4 (1.49) | 14.9 (1.45)
Statistical Analysis 1: Comparison: Lumateperone vs Placebo; Test type: Superiority; p = 0.005, ANCOVA; Least Squares Mean Difference = 4.6, 95% CI 2-sided [1.42 to 7.69]

ADVERSE EVENTS:
Time Frame: From signing ICF until end of study procedures (~10 weeks), including 6 weeks of double-blind treatment.
Arm/Group | Lumateperone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/188 | 0/189
Serious Adverse Events (participants affected / at risk) | 1/188 | 0/189
Other Adverse Events (participants affected / at risk) | 58/188 | 31/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lumateperone (N=188) | Placebo (N=189)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lumateperone (N=188) | Placebo (N=189)
Headache (Nervous system disorders) | 33 | 19
Somnolence (Nervous system disorders) | 16 | 2
Nauseau (Gastrointestinal disorders) | 12 | 4
Dizziness (Nervous system disorders) | 9 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT03249376/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/76/NCT03249376/SAP_001.pdf